CLINICAL TRIAL: NCT03613415
Title: Evaluation of Implant's Primary Stability Using Densah Bur Versus Expander in Patients With Missing Maxillary Premolar (A Randomized Clinical Trial)
Brief Title: Implant Stability Using Densah Bur Versus Expander
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hisham Mahmoud Riad, Principal Investigator (doctor), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Expansion by densah bur
Record Dates: First submitted 2018-07-23; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Missing Maxillary Premolar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: * Each patient will be given a code by the researcher (T.A.) and the observers will be blind to which group this case belong.
  * Patients, evaluators and statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expansion by Densah bur (Experimental): * Scrubbing and draping of the patient in a standard fashion for intra oral procedures followed by local anesthesia administration to the patient.
  * A mid crestal flap will be reflected.
  * For both groups the implant manufacturer's pilot drill will be used to perform a standard osteotomy of 10 mm depth.
  * Sequential use of Densah bur under copious irrigation.
  * An implant of 3.9*10 mm will be inserted.
  * Smart peg will be placed on implant and Osstell will be used to record ISQ.
  * Healing collars will be placed on implants.
  * Flap will be prepared for closure and suturing.
  Interventions: Other: Expansion
- Expander (Active Comparator): Scrubbing and draping of the patient in a standard fashion for intra oral procedures followed by local anesthesia administration to the patient.
  * A mid crestal flap will be reflected.
  * For both groups the implant manufacturer's pilot drill will be used to perform a standard osteotomy of 10 mm depth.
  * Sequential use of screw expanders.
  * An implant of 3.9*10 mm will be inserted.
  * Smart peg will be placed on implant and Osstell will be used to record ISQ.
  * Healing collars will be placed on implants.
  * Flap will be prepared for closure and suturing.
  Interventions: Other: Expansion

INTERVENTIONS:
Other: Expansion — non invasive technique to increase thickness of thin ridge

SUMMARY:
evaluating use of Densah bur in thin ridge enhance implant's primary stability when compared to screw expander.

ELIGIBILITY:
Inclusion Criteria:

* Patients with partial edentulous maxillary premolar area with crestal thickness ranging from 4 to 6 mm.
* Age 25 - 50 years.
* No intraoral soft tissue or hard tissue pathosis.
* No systemic condition contraindicating implant placement.

Exclusion Criteria:

* Ridges thickness less than 4 mm.
* Coexisting vertical defect.
* Heavy smokers (more than 20 cigarettes per day).
* Patients with systemic disease that may affect normal healing.
* Patient with psychiatric problems.
* History of radiation therapy to the head and neck region.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
implant's primary stability | intraoperative at time of surgery
  After implant placement, Implant stability will be measured by Ostell device.
implant's primary stability | Implant stability will be measured at second week
  Implant stability will be measured by Ostell device.
implant's primary stability | Implant stability will be measured at fourth week
  Implant stability will be measured by Ostell device.
implant's primary stability | Implant stability will be measured at sixth week
  Implant stability will be measured by Ostell device.
implant's primary stability | Implant stability will be measured at eighth week
  Implant stability will be measured by Ostell device.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zarb GA, Schmitt A. The longitudinal clinical effectiveness of osseointegrated dental implants: the Toronto study. Part III: Problems and complications encountered. J Prosthet Dent. 1990 Aug;64(2):185-94. doi: 10.1016/0022-3913(90)90177-e. PMID 2202818
- [Background] Branemark PI. Osseointegration and its experimental background. J Prosthet Dent. 1983 Sep;50(3):399-410. doi: 10.1016/s0022-3913(83)80101-2. No abstract available. PMID 6352924
- [Background] Branemark PI, Svensson B, van Steenberghe D. Ten-year survival rates of fixed prostheses on four or six implants ad modum Branemark in full edentulism. Clin Oral Implants Res. 1995 Dec;6(4):227-31. doi: 10.1034/j.1600-0501.1995.060405.x. PMID 8603114
- [Background] Albrektsson T, Branemark PI, Hansson HA, Lindstrom J. Osseointegrated titanium implants. Requirements for ensuring a long-lasting, direct bone-to-implant anchorage in man. Acta Orthop Scand. 1981;52(2):155-70. doi: 10.3109/17453678108991776. PMID 7246093
- [Background] Marquezan M, Osorio A, Sant'Anna E, Souza MM, Maia L. Does bone mineral density influence the primary stability of dental implants? A systematic review. Clin Oral Implants Res. 2012 Jul;23(7):767-74. doi: 10.1111/j.1600-0501.2011.02228.x. Epub 2011 Jun 2. PMID 21635560
- [Background] Trisi P, De Benedittis S, Perfetti G, Berardi D. Primary stability, insertion torque and bone density of cylindric implant ad modum Branemark: is there a relationship? An in vitro study. Clin Oral Implants Res. 2011 May;22(5):567-70. doi: 10.1111/j.1600-0501.2010.02036.x. Epub 2010 Nov 19. PMID 21087320
- [Background] Turkyilmaz I, Aksoy U, McGlumphy EA. Two alternative surgical techniques for enhancing primary implant stability in the posterior maxilla: a clinical study including bone density, insertion torque, and resonance frequency analysis data. Clin Implant Dent Relat Res. 2008 Dec;10(4):231-7. doi: 10.1111/j.1708-8208.2008.00084.x. Epub 2008 Apr 1. PMID 18384409
- [Background] Adell R, Lekholm U, Grondahl K, Branemark PI, Lindstrom J, Jacobsson M. Reconstruction of severely resorbed edentulous maxillae using osseointegrated fixtures in immediate autogenous bone grafts. Int J Oral Maxillofac Implants. 1990 Fall;5(3):233-46. PMID 2098327
- [Background] Nedir R, Bischof M, Briaux JM, Beyer S, Szmukler-Moncler S, Bernard JP. A 7-year life table analysis from a prospective study on ITI implants with special emphasis on the use of short implants. Results from a private practice. Clin Oral Implants Res. 2004 Apr;15(2):150-7. doi: 10.1111/j.1600-0501.2004.00978.x. PMID 15085870
- [Background] Urban IA, Nagursky H, Lozada JL, Nagy K. Horizontal ridge augmentation with a collagen membrane and a combination of particulated autogenous bone and anorganic bovine bone-derived mineral: a prospective case series in 25 patients. Int J Periodontics Restorative Dent. 2013 May-Jun;33(3):299-307. doi: 10.11607/prd.1407. PMID 23593623
- [Background] Menoni A, Bernardello F, Spinato S, Zaffe D. Full-arch vertical reconstruction of an extremely atrophic mandible with "box technique". A novel surgical procedure: a clinical and histologic case report. Implant Dent. 2013 Feb;22(1):2-7. doi: 10.1097/ID.0b013e318278fa1c. PMID 23287979
- [Background] Khoury, F. and Khoury, C.H., 2007. Mandibular bone block grafts: diagnosis, instrumentation, harvesting techniques and surgical procedures. In Bone augmentation in oral implantology. Quintessence, Berlin.
- [Background] Misch CM. Comparison of intraoral donor sites for onlay grafting prior to implant placement. Int J Oral Maxillofac Implants. 1997 Nov-Dec;12(6):767-76. PMID 9425757
- [Background] Simion M, Baldoni M, Zaffe D. Jawbone enlargement using immediate implant placement associated with a split-crest technique and guided tissue regeneration. Int J Periodontics Restorative Dent. 1992;12(6):462-73. PMID 1298734
- [Background] Takahashi T, Funaki K, Shintani H, Haruoka T. Use of horizontal alveolar distraction osteogenesis for implant placement in a narrow alveolar ridge: a case report. Int J Oral Maxillofac Implants. 2004 Mar-Apr;19(2):291-4. PMID 15101603
- [Background] Laurie SW, Kaban LB, Mulliken JB, Murray JE. Donor-site morbidity after harvesting rib and iliac bone. Plast Reconstr Surg. 1984 Jun;73(6):933-8. doi: 10.1097/00006534-198406000-00014. PMID 6374708
- [Background] Felice P, Pistilli R, Lizio G, Pellegrino G, Nisii A, Marchetti C. Inlay versus onlay iliac bone grafting in atrophic posterior mandible: a prospective controlled clinical trial for the comparison of two techniques. Clin Implant Dent Relat Res. 2009 Oct;11 Suppl 1:e69-82. doi: 10.1111/j.1708-8208.2009.00212.x. Epub 2009 Aug 3. PMID 19681938
- [Background] Nkenke E, Schultze-Mosgau S, Radespiel-Troger M, Kloss F, Neukam FW. Morbidity of harvesting of chin grafts: a prospective study. Clin Oral Implants Res. 2001 Oct;12(5):495-502. doi: 10.1034/j.1600-0501.2001.120510.x. PMID 11564110
- [Background] Young VL, Schuster RH, Harris LW. Intracerebral hematoma complicating split calvarial bone-graft harvesting. Plast Reconstr Surg. 1990 Oct;86(4):763-5. doi: 10.1097/00006534-199010000-00029. PMID 2217594
- [Background] Summers RB. A new concept in maxillary implant surgery: the osteotome technique. Compendium. 1994 Feb;15(2):152, 154-6, 158 passim; quiz 162. PMID 8055503
- [Background] Tatum H Jr. Maxillary and sinus implant reconstructions. Dent Clin North Am. 1986 Apr;30(2):207-29. PMID 3516738
- [Background] Demarosi F, Leghissa GC, Sardella A, Lodi G, Carrassi A. Localised maxillary ridge expansion with simultaneous implant placement: a case series. Br J Oral Maxillofac Surg. 2009 Oct;47(7):535-40. doi: 10.1016/j.bjoms.2008.11.012. Epub 2009 Jan 15. PMID 19150155
- [Background] Flanagan D. Labyrinthine concussion and positional vertigo after osteotome site preparation. Implant Dent. 2004 Jun;13(2):129-32. doi: 10.1097/01.id.0000127527.44561.b8. PMID 15179088
- [Background] Siddiqui AA, Sosovicka M. Lateral bone condensing and expansion for placement of endosseous dental implants: a new technique. J Oral Implantol. 2006;32(2):87-94. doi: 10.1563/786.1. PMID 16704111
- [Background] Cortes AR, Cortes DN. Nontraumatic bone expansion for immediate dental implant placement: an analysis of 21 cases. Implant Dent. 2010 Apr;19(2):92-7. doi: 10.1097/ID.0b013e3181d46f46. PMID 20386211
- [Background] Lee EA, Anitua E. Atraumatic ridge expansion and implant site preparation with motorized bone expanders. Pract Proced Aesthet Dent. 2006 Jan-Feb;18(1):17-22. PMID 16805345
- [Background] Nishioka RS, Souza FA. Bone spreading and standardized dilation of horizontally resorbed bone: technical considerations. Implant Dent. 2009 Apr;18(2):119-25. doi: 10.1097/ID.0b013e318198e517. PMID 19359862
- [Background] Trisi P, Berardini M, Falco A, Podaliri Vulpiani M. New Osseodensification Implant Site Preparation Method to Increase Bone Density in Low-Density Bone: In Vivo Evaluation in Sheep. Implant Dent. 2016 Feb;25(1):24-31. doi: 10.1097/ID.0000000000000358. PMID 26584202
- [Background] Trisi P, Perfetti G, Baldoni E, Berardi D, Colagiovanni M, Scogna G. Implant micromotion is related to peak insertion torque and bone density. Clin Oral Implants Res. 2009 May;20(5):467-71. doi: 10.1111/j.1600-0501.2008.01679.x. PMID 19522976
- [Background] Todisco M, Trisi P. Bone mineral density and bone histomorphometry are statistically related. Int J Oral Maxillofac Implants. 2005 Nov-Dec;20(6):898-904. PMID 16392347
- [Background] Huwais S, Meyer EG. A Novel Osseous Densification Approach in Implant Osteotomy Preparation to Increase Biomechanical Primary Stability, Bone Mineral Density, and Bone-to-Implant Contact. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):27-36. doi: 10.11607/jomi.4817. Epub 2016 Oct 14. PMID 27741329
- [Background] Lahens B, Neiva R, Tovar N, Alifarag AM, Jimbo R, Bonfante EA, Bowers MM, Cuppini M, Freitas H, Witek L, Coelho PG. Biomechanical and histologic basis of osseodensification drilling for endosteal implant placement in low density bone. An experimental study in sheep. J Mech Behav Biomed Mater. 2016 Oct;63:56-65. doi: 10.1016/j.jmbbm.2016.06.007. Epub 2016 Jun 10. PMID 27341291